CLINICAL TRIAL: NCT05342857
Title: Investigation of the Maximal Treatment Interval and Long-term Remission and the Associated Factors of Neovascular AMD Treated With Anti-VEGF Using Treat and Extend Strategy
Brief Title: Maximum Treatment Interval With Aflibercept T&E
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20211006R
Record Dates: First submitted 2022-04-05; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Aflibercept Injection [Eylea] — Aflibercept 2.0 mg with the T&E criteria in Taiwan local consensus

SUMMARY:
To evaluate the duration of effectiveness of anti-VEGF (Aflibercept) by analyzing the percentage of patients whose maximum treatment interval is extended to 16 weeks and beyond in 24 months and their long-term remission.

DETAILED DESCRIPTION:
This is an Observational, prospective, single arm study. The distribution of maximum treatment interval extended within 2 year among nAMD patients with Aflibercept Treat-and-Extend(T&E) regimen will be analyzed. And Clinical indicators for fast extension of treatment interval and emering disease activity will be captured.

To maximize Vision acuity (VA) outcome and reduce treatment burden of neovascular age-related macular degeneration (nAMD) patients, the T&E regimen has become popular in recent years. Sufficient drug durability is the key element to support T&E regimen. Clinical trials with aflibercept suggest a longer duration of VEGF suppression than with bevacizumab or ranibizumab, which is also supported by pharmacokinetic models, and mean duration of vitreous VEGF suppression by aflibercept injection was demonstrated as > 71 ± 18 days. With these attributes, while managed by intravitreal injection aflibercept (IVI-ALF) T&E regimen, it has been shown in ALTAIR study that around 40% and 60% of patients had treatment interval extended to 12 week and 16 weeks at week 96 respectively.

Nevertheless, it was observed that the distribution of treatment interval is polarized, a group of patients would eventually reach a stable disease status with only few treatments needed per year, while another group of patients may still need more intensive treatment even shorter than 8 week interval. To maximize benefit of patients with practical and personalized IVT-AFL T&E regimens, it is important to provided further evidence to support maximizing treatment interval as well as clinical indicators to take precise action to active disease. Therefore, this study is designed to understand the potential durability of Aflibercept by analyzing maximum treatment interval with IVT-AFL in 2 years, and explore clinical indicators to guide optimal T&E regimen for each patient.

Patients are treated with Aflibercept 2.0 mg following the T&E criteria in Taiwan local consensus (listed as below). Once the treatment interval is extended to 16 weeks, and the patient has two consecutive 16-week treatment interval, treatment strategy will be changed to pro re nata (PRN) with monthly follow-up. IVI-AFL will immediately be applied once there is any disease activity detected.

During the study, patients will be monitored with BCVA, fundus photograph, structural OCT, OCT Angiography.

T&E criteria in Taiwan local consensus:

* Extension: No BCVA loss ≥ 5 ETDRS letters (or 1 line of Snellen chart) AND dry retina§,†, #
* Maintain: No BCVA loss ≥ 5 ETDRS letters (or 1 line of Snellen chart) AND non-increased fluid§
* Shortening: Any increased fluid with BCVA loss ≥ 5 ETDRS letters (or 1 line of Snellen chart)‡, # OR new macular hemorrhage OR new neovascularization

"§"Absence of macular hemorrhage and neovascularization is required.

"†"Non-increased fluid after 3 more consecutive monthly injections following initial treatment could be considered as persistent fluid, and the injection interval could be extended if VA is stable.

"‡" Either increased fluid or BCVA loss ≥ 5 ETDRS letters alone could be maintained at current treatment interval.

"#" Extension or shortening can be by 2 or 4 weeks

ELIGIBILITY:
Inclusion Criteria:

* -Treatment-naïve patients with subfoveal CNV secondary to wet AMD and PCV, with visual impairment being exclusively due to an symptomatic neovascular AMD.
* - -Clinical status meet the national reimbursement criteria

Exclusion Criteria:

* - Any contraindications as listed in the local intravitreal aflibercept package insert
* - Any active periocular or ocular infection or inflammation at baseline
* - Uncontrolled glaucoma (intraocular pressure [IOP] ≥30 mm Hg on medication) at baseline
* - Neovascularisation of the iris or neovascular glaucoma at baseline
* - Visually significant cataract, severe vitreous haemorrhage, rhegmatogenous retinal detachment, proliferative diabetic retinopathy or CNV of any cause other than wet AMD at baseline
* - Structural damage to the center of the macula in either eye that is likely to preclude improvement in VA following the resolution of macular edema or any other condition expected to permanently limit VA outcomes over the course of the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Treatment-naïve nAMD and PCV patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients whose maximum treatment interval is extended to 24 months | 2 years

SECONDARY OUTCOMES:
Find the prediction factors associated with extension to 16 weeks and beyond by univariate and multivariate analysis | 2 years
Find the prediction factors associated with occurrence of disease activity by univariate and multivariate analysis | 2 years
The percentage of patients whose maximum treatment interval is extended to 16 weeks and beyond in 24 months in PCV and wAMD subgroup | 2 years
Mean change in BCVA from baseline to month 24 | 2 years
Mean change in central subfield thickness from baseline to month 24 | 2 years
Proportion of patients who gain ≧15 ETDRS letters from baseline to month 24 | 2 years
Mean number of injections in each group from baseline to month 24 | 2 years
Mean treatment interval from baseline to month 24 | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shin Kong Memorial Wu Ho-Su Hospital, Taipei, Taiwan